CLINICAL TRIAL: NCT06386809
Title: Investigation of the Effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation in Bruxism- Randomised Controlled Single Blinded Study
Brief Title: Effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation in Bruxism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024 -25
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Bruxism
Keywords: bruxism; vagus; stimulation; parasympathetic
MeSH Terms: conditions — Bruxism | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVNS group (Experimental)
  Interventions: Device: TAVNS; Other: Exercise program
- Exercise group (Other)
  Interventions: Other: Exercise program

INTERVENTIONS:
Device: TAVNS — TAVNS is a recently introduced treatment involving transcutaneous electrical stimulation of the auricular branch of the vagus nerve with VAGUSTIM device.
  Arms: TAVNS group
Other: Exercise program — Rocabado 6x6 exercises will be applied in our study. Rocabado exercise, which is the most commonly used exercise method in the literature, is a set of exercises for the craniocervical and craniomandibular system.

SUMMARY:
Our study aimed to investigate the effects of transcutaneous auricular vagus nerve stimulation (TAVNS) application on treatment efficacy in bruxism in terms of masseter muscle activity, pain, stress level, sleep and life quality, and autonomic functions.

DETAILED DESCRIPTION:
Our study was designed as a randomized, single-blind experimental clinical trial. It was planned to include 40 individuals diagnosed with bruxism in our research. Outcome measurements and assessments will be performed immediately after the participants are recruited and at the end of the 8-week program. Pain intensity, oral health quality of life, stress level and sleep quality will be assessed by self-report through questionnaires. Pressure pain threshold and muscle activation for the masseter muscle and heart rate variables measurements will be performed by physiotherapists. After completing the initial evaluations, the participants will be randomly divided into two groups. An eight-week exercise program will be applied to the control group. In the TAVNS group, in addition to the eight-week exercise program, TAVNS will be used twice weekly for 16 sessions with the VAGUSTIM device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bruxism between the ages of 18-65,
* A history of bruxism for at least 6 months,
* Individuals with masseter muscle pain GAS≥4 at rest and during mastication

Exclusion Criteria:

* Masseter botox application in the last 6 months,
* Regular use of analgesics and anti-inflammatories that affect the OSS,
* Presence of infection or tumoral structures within intraoral structures,
* Wearing multiple ear piercings,
* With TMJ disc displacement and joint degeneration,
* Musculoskeletal problem with evidence of cervical or TMJ fracture, systemic disease, specific pathologic condition,
* Any surgical operation related to a cervical or TMJ problem,
* Less than 6 months of cervical or TMJ-related physiotherapy and rehabilitation services,
* The one with facial paralysis,
* Diagnosed psychiatric illness

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | 8 weeks
  Participants' pain intensity will be assessed using the Visual Analog Scale, is a simple, reliable and short-term method commonly used in the clinic to measure pain intensity.The participant is told that the most severe pain he/she experiences is 10, and if he/she has no pain, the pain intensity is 0. The participant will be asked to mark a number between 0 and 10 corresponding to the intensity of pain in the masticatory muscles at rest and during chewing.
Oral Health Quality of Life | 8 weeks
  The Oral Health Impact Profile is revised to comprehensively measure the discomfort, disability and handicap related to oral and dental health. The scale consists of 14 questions in 7 dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. The lowest score that can be obtained from the scale is 0, while the highest score that can be obtained is 56. A high score indicates poor quality of life.
Stress Level | 8 weeks
  The Perceived Stress Scale-14 is a self-report scale designed to assess one's perception of the degree to which a particular situation in daily life is considered stressful. It consists of 14 items and is rated on a 4-point Likert scale ('0: never' to '4: very often'). A high total score indicates a high level of perceived stress.
Sleep Quality | 8 weeks
  Pittsburgh Sleep Quality Index will be used to assess the sleep quality of the participants. It assesses sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime work disturbance and sleep latency and consists of a total of 24 questions. The total score ranges from 0-21, with 5 and above indicating "poor sleep quality".
Pressure Pain Threshold | 8 weeks
  In our study, pressure pain threshold measurement of the dominant and non-dominant side masseter muscle before and after activity will be evaluated with Baseline manual algometer (2.5 kg-11 lb).
Muscle Activation Measurement | 8 weeks
  In our study, four-channel 'Neurotrac Myoplus Pro 4 EMG Biofeedback' device will be used for superficial EMG measurements. The EMG work-rest mode of the device will be used in the measurement and the masseter muscle activation during contraction and relaxation will be measured by asking the participant to clench his/her teeth 5 times consecutively, 5 seconds contraction time, 5 seconds relaxation time. Neurotrac PC Software program will be used for electromyographic analysis during the measurement.
Measurement of heart rate variability/ Autonomic nervous system evaluation | 8 weeks
  All participants included in the study will undergo a 5-minute heart rate variability measurement test with the Polar H10 chest strap device. The data obtained after the measurement will be analyzed with Kubios program. Stress index (cardiovascular system stress), PNS index (parasympathetic nervous system dominance), SNS index (sympathetic nervous system dominance), LF power (sympathetic activity) and HF power (parasympathetic activity) parameters will be recorded in Kubios program.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey (Türkiye)

REFERENCES:
- [Derived] Guzel HC, Turkmen OB, Mutlu EK, Turkmen G, Sakar O, Ormeci GO. Effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation in Bruxism: A Randomised, Controlled, Single-Blind Experimental Trial. J Oral Rehabil. 2026 Feb;53(2):493-504. doi: 10.1111/joor.70096. Epub 2025 Nov 10. PMID 41211817